CLINICAL TRIAL: NCT06106321
Title: Transalveolar Crest Parietal Sinus Floor Lift and Secondary Lift for Postoperative Improvement of Neonatal Bone Mass in Sinus: a Prospective Clinical Study in the Posterior Maxillary Region
Brief Title: Primary and Secondary Elevations of Maxillary Sinuses: a Prospective Clinical Study in the Posterior Maxillary Region
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2023-358
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Tooth Loss
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transalveolar crest parietal maxillary sinus floor secondary lift (Experimental): In order to achieve minimally invasive surgery (RBH≤5mm) in patients with severe deficiency of residual bone height in the posterior maxillary region and obtain reliable clinical research results, a secondary sinus floor lifting technique combining the advantages of maxillary sinus lift with the low risk of maxillary sinus lift is proposed.
  Interventions: Procedure: transalveolar crest parietal maxillary sinus floor secondary lift
- Transalveolar crest parietal maxillary sinus floor lift (Active Comparator): Transalveolar crest parietal maxillary sinus floor lift (OSFE) requires a residual bone height of at least 5 mm and implant placement at the same time. Its advantages are simple operation, shorter surgical time, reduced trauma and reduced postoperative complications, and the concept of minimally invasive implant surgery is reflected in OSFE.
  Interventions: Procedure: Transalveolar crest maxillary sinus floor lift

INTERVENTIONS:
Procedure: Transalveolar crest maxillary sinus floor lift — Transalveolar crest maxillary sinus floor lift + bone grafting + implant implant is used
  Arms: Transalveolar crest parietal maxillary sinus floor lift
Procedure: transalveolar crest parietal maxillary sinus floor secondary lift — Transalveolar crest parietal maxillary sinus floor secondary lift + bone grafting + implant implantation were used body
  Arms: Transalveolar crest parietal maxillary sinus floor secondary lift

SUMMARY:
About 40 people will participate in the study, which will be conducted at Southern Medical University Southern Hospital. All subjects need to sign an informed consent form before screening, and successful subjects can enter the study. Experimental and control subjects were treated according to the protocol. Treatment was held until the participant entered a follow-up period, or until any of the withdrawal criteria were met. According to conventional clinical practice, the study needs to evaluate the patient's subjective perception and soft and hard tissue changes at 3 months, 6 months, and 1 year after successful implant placement. The specific process is divided into: 1. Screening period: All subjects need to complete the relevant examinations of the screening period before enrollment, and screen according to the admission criteria. (1) Sign informed consent; (2) Record demographic data: date of birth, gender, initials; (3) Medical history and physical examination: collection includes understanding of any current or past diseases, medications, drug allergy history, surgical history, radiotherapy and chemotherapy history, ethnic background, smoking history, whether alcoholism, oral hygiene habits and oral examination, etc.; (4) Among them, oral examination includes the whole oral health before and after surgery and oral and maxillofacial CBCT imaging examination; 2. Treatment period: the control group underwent transalveolar crest parietal maxillary sinus floor lift immediately after implants; The experimental group underwent implant implantation after 6 months of transalveolar crest parietal maxillary sinus floor lift. 3. Follow-up period: The study needs to evaluate the subjective feelings and soft and hard tissue changes of patients at 3 months, 6 months and 1 year after implant placement.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥ 18 years old
2. If the posterior maxillary tooth is missing for ≥ 3 months, the patient requires implant restoration and the preoperative examination meets the indications for intramaxillary sinus lift
3. Can be scanned with radiology equipment before and after surgery
4. RBH ≤ 5mm, alveolar ridge width ≥5mm, each implant site is measured on CBCT
5. During implant healing, there is no removable restoration at the implant site
6. No history of acute or chronic sinusitis disease, no history of maxillary sinus disease, and no history of previous maxillary sinus surgery
7. Be willing to sign informed consent and authorization form, and be able to return to the clinic on time

Exclusion Criteria:

1. Heavy smokers (10 cigarettes smoked ≥ day)
2. Uncontrolled diabetes (glycated hemoglobin >7%), metabolic bone disease, autoimmune disease or other systemic diseases, the body can hardly withstand implant surgery
3. Mentally unable, pregnant or pregnant women
4. Any history of contraindications or significant impact on dental implant placement, such as bisphosphonate drug use, chemotherapy or immunosuppressants, head and neck radiotherapy, autoimmune disease, and hypertension
5. Untreated periodontal disease, endodontics, or other oral diseases
6. Bruxism patients
7. Previous implant implant failure at the surgical site
8. Anatomical changes in the maxillary sinus, such as maxillary sinus septum or mucosal swelling (defined as the mean thickness of the Schneider membrane at the base of the maxillary sinus > 2 mm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-07 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Neonatal bone mass in the sinus | 3, 6, 12 months after implantation
  The sum of bone mass (ABH) in the apical region and the elevation height (IPL) of the maxillary sinus floor (IPL) was measured by CBCT 3, 6, and 12 months after implantation

SECONDARY OUTCOMES:
Remaining alveolar ridge height | Preoperatively, 3, 6, 12 months after implantation
  CBCT was used to measure the distance from the lowest coronal level of bone-implant contact to the apical level of bone-implant contact with sinus floor cortical bone
Maxillary sinus floor elevation height | 3, 6, 12 months after implantation
  3 months, 6 months, and 1 year after implantation, CBCT was used to measure the distance from the root tip of the implant to the cortical line of the sinus floor
Peri-implant marginal bone resorption | Preoperatively, 3, 6, 12 months after implantation
  CBCT was used to measure the difference between marginal bone level and marginal bone level baseline before surgery, 3 months, 6 months, and 1 year after implantation

CONTACTS AND LOCATIONS:
Locations (1):
- NanFang Hospital of Sourthern Medical University, Guangzhou, Guangdong, China